# Statistical Analysis Plan (SAP)

Evaluation of Tc 99m Tilmanocept Imaging for the Early Prediction of Anti-TNFα Therapy Response in Patients with Moderate to Severe Active Rheumatoid Arthritis (RA)

Study No: NAV3-33

Version 4.0

October 6, 2023

Prepared for Navidea Biopharmaceuticals, Inc. 4995 Bradenton Avenue, Suite 240 Dublin, OH 43017

Prepared by STATKING Clinical Services 3570 Pleasant Ave Hamilton, OH 45015 513-858-2989

www.statkingclinical.com



# **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

I agree to the format and content of this document.

| Approved by: Michael S. Blue, MD Chief Medical Officer Navidea Biopharmaceuticals 4995 Bradenton Avenue, Suite 240 Dublin, Ohio 43017 mblue@navidea.com | 10 10 23<br>Date |
|---|---|
| Authored by: Zachary Steckler, MS Statistician STATKING Clinical Services 3570 Pleasant Ave Hamilton, OH 45015 zachary@gd3services.com | 10/10/2023<br>Date |
| Approved by (internal review): Lear Services Ian Lees, MS Statistician STATKING Clinical Services 3570 Pleasant Ave Hamilton, OH 45015 ilees@gd3services.com | 10 10 7023<br>Date |

Approved by:

Clare Gerger

10-10-2023

Date

Clare Geiger, RN
Project Manager
STATKING Clinical Services
3570 Pleasant Ave
Hamilton, OH 45015
cgeiger@gd3services.com

# **Revision History**

#### Version 3.0 to 4.0

- Updated signature page to reflect changes in staff and contacts
- Removed non-bucketing algorithms, so that all subjects with TUV<sub>global[b]</sub> <</li>
   5 will be predicted non-responders
- Clarified secondary objective in section 1.0 for qualitative assessment of Tc 99m tilmanocept imaging by removing language pertaining to change from baseline
- Added description of tipping point analyses for mean imputation of clinical status at week 24 and TUV prediction to section 2.3
- Modified section 4.1.4 to indicate that the secondary efficacy variables will be based on bucketing algorithms
- Removed table and listing shells for non-bucketing algorithms
- Removed columns, footnotes, and annotations in TLF shells for nonbucketing algorithms
- Added figures to summarize tipping point analyses using 95% confidence intervals to TLF shells

#### Version 2.0 to 3.0

- Added description of analysis of qualitative assessments to section 4.2.3
- Added description of analysis of the additive effect of either quantitative or qualitative assessment of Tc 99m tilmanocept imaging to section 4.2.3
- Modified description of concordance of improvement classification of each algorithm with clinical improvement criteria to indicate that p-values for sensitivity and specificity will be included
- Added tables for concordance of qualitative assessment of Tc 99m tilmanocept imaging with clinical improvement criteria
- Added tables for concordance of qualitative plus quantitative assessment of Tc 99m tilmanocept imaging with clinical improvement criteria
- Added tables for summary of generalized linear mixed model to asses the additive effect of either quantitative or qualitative assessment of Tc 99m tilmanocept imaging on patient response status
- Added p-values for all clinical assessments in addition to those for ACR50 to tables 15-22
- Added data listing for qualitative imaging assessments
- Added data listing for qualitative plus quantitative assessments which differ from original quantitative assessment
- Updated TLF table of contents to remove redundant tables
- Added new tables and listings to TLF table of contents
- Renumbered TLFs to include new additions

#### **Version 1.0 to 2.0**

- Changed intent-to-diagnose population in section 2.2 to include all subjects who were injected with Tc 99m tilmanocept at visit 2 and received planar imaging of the hands at visit 2, regardless of if they received any other assessments.
- Changed wording in section 1.3 to specify that at least the same two of three readers must reject both null hypotheses for the two co-primary endpoints to be achieved.
- Added detail in section 2.3 regarding imputation strategies, and proposed secondary imputation strategy for some missing data scenarios if primary imputation strategy does not work.
- Added detail in section 4.1.1.1 regarding the possibility for a patient's TUV prediction from bucketing vs. non-bucketing to differ, and how these findings will be summarized.
- Added tables 27-28 to summarize the number of patients who TUV predictions from bucketing vs. non-bucketing differ.
- Added data listing 28 to provide detail on patients who TUV predictions from bucketing vs. non-bucketing differ.

# **Table of Contents**

| APPROVAL PAGE | 2 |
|------------------------------------------------------|----|
| REVISION HISTORY | 4 |
| LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 8 |
| INTRODUCTION | 10 |
| 1.0 SYNOPSIS OF STUDY DESIGN/PROCEDURES | 10 |
| 1.1 Design and Treatment | 12 |
| 1.2 Study Procedures | 12 |
| 1.3 Sample Size | 13 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 15 |
| 2.1 Types of Analyses | 15 |
| 2.2 Analysis Populations | 15 |
| 2.2.1 Subgroup Definitions and Considerations | 16 |
| 2.3 Missing Data Conventions | 16 |
| 2.4 Interim Analyses | 17 |
| 2.5 Calculation of TUV | 17 |
| 2.6 Study Center Considerations in the Data Analysis | 19 |
| 2.7 Documentation and Other Considerations | 19 |
| 3.0 ANALYSIS OF BASELINE PATIENT CHARACTERISTICS | 19 |
| 4.0 ANALYSIS OF EFFICACY | 19 |
| 4.1 DESCRIPTION OF EFFICACY VARIABLES | 19 |
| 4.1.1 Definition of Responder/Non-Responder Status | 19 |
| 4.1.1.1 Prediction Algorithms | 19 |

| 4.1.1.2 Clinical Assessments | 20 |
|---------------------------------------------------------|----|
| 4.1.2 Description of Primary Efficacy Variables | 21 |
| 4.1.3 Description of Key Secondary Efficacy Variables | 21 |
| 4.1.4 Description of Secondary Efficacy Variables | 22 |
| 4.2 Analysis of Efficacy Variables | 23 |
| 4.2.1 Analysis of Primary Efficacy Variables | 23 |
| 4.2.2 Analysis of Key Secondary Efficacy Variables | 24 |
| 4.2.3 Analysis of Secondary Efficacy Variables | 24 |
| 5.0 ANALYSIS OF SAFETY | 26 |
| 6.0 OTHER RELEVANT DATA ANALYSES/SUMMARIES | 27 |
| 6.1 Patient Completion | 27 |
| 6.2 Physical Exam | 27 |
| 6.3 Study Drug Administration | 28 |
| 6.4 RA Evaluation and Screening Physical Exam | 28 |
| 6.5 Concomitant Medications | 28 |
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 29 |
| 8.0 REFERENCES | 33 |
| APPENDIX A – TABLES, FIGURES AND LISTING SPECIFICATIONS | 34 |
| APPENDIX B – TABLE. FIGURE. AND LISTING SHELLS | 36 |

# **List of Abbreviations and Definitions of Terms**

| Term | Definition |
|---|---|
| Δ | Greek letter delta, used to represent the change in a particular |
| | variable |
| μg | microgram |
| ACPA | anti-citrullinated protein/peptide antibody |
| ACR/EULAR | American College of Rheumatology/ European League |
| | Against Rheumatism |
| AE | adverse event |
| Anti-TNF-α | Anti-Tumor Necrosis Factor $\alpha$ biological Disease Modifying |
| bDMARD | Anti-Rheumatic Drug |
| CDAI | Clinical Disease Activity Index |
| CFB | change from baseline |
| CI | confidence interval |
| CRF | case report form |
| СТ | X-ray computed tomography |
| DAS28 | Disease activity score used with the ACR/EULAR 2010 RA |
| | guidelines |
| ECG | electrocardiogram |
| FDA | Food and Drug Administration |
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| HC(s) | healthy control(s) |
| ICH | International Conference on Harmonization |
| ITD | intent-to-diagnose |
| IV | intravenous |
| mCi | milliCurie (37x10 <sup>6</sup> becquerels; 37megabecquerels) |
| MCP | metacarpophalangeal |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | macrophage-involved contribution |
| NPV | Negative Predictive Value |
| OA | Overall Accuracy |
| PIP | proximal interphalangeal |
| PP | per protocol |
| PPV | Positive Predictive Value |
| PR | the time from the onset of the P wave to the start of the QRS |
| | complex |
| QRS | time from the start of the Q wave to the end of the S wave, |
| | representing ventricular depolarization |
| QT | time from the start of the Q wave to the end of the T wave |
| QTcF | QT interval with Fridericia's correction formula |
| RA | rheumatoid arthritis |
| ROI | region of interest |
| SAE | serious adverse event |

| Term | Definition |
|-------------|---------------------------------------------------------------|
| SAP | statistical analysis plan |
| SJC | swollen joint count |
| SOC | system organ class |
| SPECT | single photon emission computed tomography |
| Tc 99m | technetium-99m metastable isotope; γ-emitting (half-life 6.02 |
| | h) |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| tilmanocept | DTPA Mannosyl Dextran (the US Adopted Name for the drug |
| | substance of Lymphoseek) |
| TJC | tender joint count |
| TUV | Tilmanocept uptake value |
| US | United States |
| WPI | Widespread Pain Index |

#### INTRODUCTION

## Description

This statistical analysis plan (SAP) is consistent with Amendment #3 of the study protocol (dated 29 September 2023) and includes details of efficacy and safety summaries for use in support of the planned trial, as outlined in ICH E3 (Structure and Content of Clinical Study Reports) and ICH E9 (Statistical Principles for Clinical Trials). Considerations were also given to the FDA Guidance for industry on Developing Medical Imaging Drug and Biological Products Part 3: Design, Analysis, and Interpretation of Clinical Studies (June 2004), FDA Guidance for Industry on Clinical Trial Imaging Endpoint Process Standards (April 2018) and Statistical Guidance on Reporting Results from Studies Evaluating Diagnostic Tests - Guidance for Industry and FDA Staff (March 2007). The study design and analysis plans align with recommendations received from the US FDA at the End of Phase 2 meeting on 01 September 2021 (IND 132943).

# 1.0 Synopsis of Study Design/Procedures

This is a prospective, multicenter, open-label study designed to evaluate the early predictive capacity of quantitative Tc 99m tilmanocept planar imaging for downstream clinical response(s) in individuals with moderate to severe rheumatoid arthritis (RA) who are candidates for change in anti-TNF $\alpha$  therapy. Temporal changes (from baseline to 5-weeks) in quantitative imaging will be correlated with longitudinal changes (from baseline to 12 weeks and baseline to 24 weeks) in RA clinical assessments, with the intent of evaluating the clinical utility of Tc 99m tilmanocept for the expedited evaluation of antirheumatic treatment efficacy when compared with longitudinal assessments in clinical practice.

The study objectives are as follows:

## **Primary:**

- To demonstrate that global tilmanocept uptake values (TUV<sub>global</sub>) obtained before initiation of anti-TNFa therapy (TUV<sub>global[b]</sub>) and at 5 weeks ± 1 week following change in therapy (TUV<sub>global[5w]</sub>) has a specificity of greater than 80% to correctly specify a clinical non-response to therapy at 24 weeks.
- To demonstrate that TUV<sub>global</sub> obtained before initiation of anti-TNFα therapy and at 5 weeks ± 1 week following change in therapy has a sensitivity of greater than 65% to correctly classify a positive clinical response to therapy at 24 weeks.

## **Key Secondary**

• To evaluate the negative predictive value (NPV) of TUV<sub>global</sub> obtained before initiation of anti-TNFα therapy (TUV<sub>global[b]</sub>) relative to a clinical non-response to therapy at 24 weeks.

## **Secondary**

- To evaluate the sensitivity and specificity of TUV<sub>global</sub> obtained before initiation of anti-TNFα therapy and at 5 weeks ± 1 week following change in therapy relative to a positive clinical response or a non-response to therapy at 12 weeks.
- To evaluate the NPV of TUV<sub>global[b]</sub> relative to a clinical non-response to therapy at 12 weeks.
- To evaluate the positive predictive value (PPV), NPV, and overall accuracy (OA) of TUV<sub>global</sub> obtained before initiation of anti-TNFα therapy and at 5 weeks ± 1 week (ΔTUVglobal<sub>[5w]</sub>) following change in therapy relative to a positive clinical response or a non-response to therapy at 12 and/or 24 weeks.
- To evaluate the qualitative assessment of Tc 99m tilmanocept imaging to predict clinical response or non-response following a change in anti-TNFα therapy.
- To evaluate the additive effect of either quantitative or qualitative assessment of Tc 99m tilmanocept imaging to the other at baseline and change from baseline to 5 weeks ± 1 week to predict clinical response or non-response following a change in anti-TNFα therapy.
- To evaluate the correlation of changes in TUV<sub>global</sub> obtained before initiation of anti-TNFα therapy and at 5 weeks ± 1 week following a change in therapy with changes in composite clinical assessments and their constituent parameters at 12 and/or 24 weeks.
- To evaluate the correlation of changes in  $TUV_{global}$  obtained before initiation of anti-TNF $\alpha$  therapy and at 5 weeks  $\pm$  1 week following a change in therapy with changes in clinical assessments at 12 and/or 24 weeks for specific anti-TNF $\alpha$  bDMARD agents.
- To evaluate the ability of changes in TUV<sub>global</sub> obtained before initiation of anti-TNFα therapy and at 12 weeks ± 1 week following change in therapy to accurately predict a clinical response or non-response at 24 weeks.
- To evaluate the correlation of changes with TUV<sub>global</sub> and changes in clinical RA assessments as a means to monitor therapy.
- To evaluate sensitivity and specificity in patient subgroups.

 To evaluate the safety of IV-administered tilmanocept radiolabeled with Tc 99m.

The statistical endpoints that address these objectives are defined in Section 4 (efficacy) and Section 5 (safety). Refer to Section 2.2.1 for subgroup definitions and considerations.

## 1.1 Design and Treatment

This is a prospective, open-label, multicenter study designed to evaluate the early predictive capacity of quantitative Tc 99m tilmanocept planar imaging for downstream clinical response(s) in individuals with moderate to severe RA who are candidates for change in anti-TNF $\alpha$  therapy.

All patients will receive an IV dose of 150 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m prior to imaging.

## 1.2 Study Procedures

Prior to the initiation of a new anti-TNF $\alpha$  therapy, patients will undergo baseline rheumatological evaluations of ACR/EULAR 2010, Clinical Disease Activity Index (CDAI), DAS28, and Health Assessment Questionnaire Disability Index (HAQ-DI) for the characterization of disease activity. After these evaluations, patients will receive an IV dose of 150 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m and undergo baseline planar imaging of the bilateral hands and wrists. Upon completion of baseline imaging procedures, patients will commence a new anti-TNF $\alpha$  bDMARD treatment regimen and return to the clinic 5 +/- 1 weeks, 12 +/- 1 weeks, and 24 +/- 1 weeks later for a series of rheumatological evaluations (including CDAI, DAS28, ACR Response Criteria, and HAQ-DI), drug administration, and bilateral hand/wrist imaging.

Images will undergo centralized quantification for the derivation of joint-specific and global TUV. At the joint level, TUV is defined as the intrapatient ratio of the average pixel intensity of a joint to the average pixel intensity of the reference region. TUV<sub>global</sub> is a per patient summary of TUV<sub>joint</sub> values greater than the normative database representing RA-specific inflammation.

All images will be read by three nuclear medicine specialists trained in the reading of these images. Each reader will work independently of the other readers. Each reader will provide both a qualitative read and map regions of interest for calculation of TUV.

Temporal differences in  $TUV_{global}$  from baseline to 5 +/- 1 weeks of therapy  $(\Delta TUV_{global[5w]})$  will be compared with longitudinal clinical outcomes at 12 +/- 1

and 24 +/- 1 weeks of therapy defined by changes in CDAI ( $\Delta$ CDAI<sub>[12/24w]</sub>), changes in ACR Response Criteria ( $\Delta$ ACR<sub>[12/24w]</sub>), and changes in DAS28 ( $\Delta$ DAS28<sub>[12/24w]</sub>) to evaluate the efficacy of TUV<sub>global</sub> for the accelerated prediction of clinical response to antirheumatic drugs.

Refer to the clinical study protocol for further details on the study procedures and for the schedule of events table.

## 1.3 Sample Size

NAV3-33 is sized with respect to achieving specified goals in the co-primary endpoints of sensitivity and specificity of  $\Delta TUV_{global[5w]}$  with bucketing. Sensitivity and specificity require knowledge of the patient's clinical status at Week 24, and so hypothesis testing will be performed after classification. The value of  $\Delta TUV_{global[5w]}$  necessary to predict response vs. non-response and the value of  $TUV_{global[5w]}$  at baseline necessary to predict non-response will be determined in advance. The classification procedure occurs in two stages, following the baseline image acquisition and (possibly) following the 5 week image acquisition and calculation of  $\Delta TUV_{global[5w]}$ . After the baseline imaging, patients whose  $TUV_{global[5w]}$  is < 5 are predicted to be non-responders. After  $\Delta TUV_{global[5w]}$  is available, patients whose  $TUV_{global[b]}$  is  $\leq 5$  and D% is  $\leq -10\%$  are predicted to be responders. All other patients are predicted to be non-responders. The Week 24 ACR50 will be used as the primary determination of clinical response for the reference standard

The hypotheses for the co-primary endpoints to be tested are:

$$H_{O1}$$
:  $\pi_{Sp} \le 0.8$   
 $H_{A1}$ :  $\pi_{Sp} > 0.8$ ;

And

$$H_{O2}$$
:  $\pi_{Se} \le 0.65$   
 $H_{A2}$ :  $\pi_{Se} > 0.65$ .

In the above  $\pi_{Sp}$  represents the true specificity of the classification procedure and  $\pi_{Se}$  represents the true sensitivity of the classification procedure when used to predict the outcome of the anti-TNF $\alpha$  bDMARD inhibitor therapy at 24 weeks. An overall two-tailed Type I error rate of 0.05 (one-tailed 0.025) was used without adjusting for multiple endpoints, as both co-primary endpoints must be achieved in order to have a successful study. If the actual specificity is 0.92 and the actual sensitivity is 0.8, and if an exact binomial test is used to test the above hypotheses, a total of 98 clinical non-responders and 100 clinical responders are

needed for 90% power of the individual tests. That is, a minimum of 198 total patients is needed. This applies to a single reader.

To evaluate the power characteristics of this process with 3 correlated readers where at least the same two of the three readers must reject both null hypotheses above, a simulation study was performed. Correlated binomial random variables were generated using a copula. The hypotheses were tested for each simulated reader using an exact binomial test, and the number of iterations where at least the same two of the three readers rejected both hypotheses was counted. Under the conditions above this procedure has power 0.93 when  $\rho=0.7$  and 0.89 when  $\rho=0.9$ .

In Arm 3 of the NAV3-31 study a ratio of 5 non-responders to 1 responder was observed. If this ratio is maintained in NAV3-33 for the  $\Delta TUV_{global[5w]}$  with bucketing predictions, a total of 600 patients is needed to achieve the desired power. That is, a total of 500 clinical non-responder patients is expected to be enrolled before reaching the required 100 clinical responders.

Taking into account a 10% dropout rate, the anticipated total sample size for the study is approximately 672 patients (560 clinical non-responders and 112 clinical responders). That is:

- Clinical Non-Responders: 90% completion rate relative to 560 enrolled patients will result in 500 completed patients
- Clinical Responders: 90% completion rate relative to 112 enrolled patients will result in 100 completed patients

Because there is uncertainty about how responding and non-responding patients will enroll, enrollment may continue until at least 560 clinical non-responders and 112 clinical responders are participating in the study. The cumulative enrollment of clinical non-responders and responders will be tracked throughout the study in order to stop enrollment once the required number has been reached for each clinical category. This tracking of clinical response and non-response status will be performed by individuals without knowledge of the TUV data. At the Sponsor's discretion, the week 12 clinical response outcomes may be used to help track enrollment.

If the two co-primary endpoints are achieved (i.e., both null hypotheses are rejected for at least the same 2 out of 3 readers), then the following hypotheses will be tested at one-tailed 0.025 for the key secondary endpoint of NPV of TUV<sub>global[b]</sub> with respect to ACR50 at week 24:

$$H_{O3}$$
:  $\pi_{NPV} \le 0.7$   
 $H_{A3}$ :  $\pi_{NPV} > 0.7$ ;

If the actual NPV is 0.85, and if an exact binomial test is used to test the above hypotheses, a total of 89 predicted non-responders using TUV<sub>global[b]</sub> are needed for 90% power and a total of 71 non-responders using TUV<sub>global[b]</sub> are needed for 80% power. Enrollment of predicted non-responders at baseline will be tracked in order to ensure enough subjects are enrolled to achieve at least 80% power for this endpoint.

All enrollment tracking will be done in aggregate by individuals without knowledge of the subject-level data. Enrollment tracking will include the total number of predicted non-responders at baseline, the total number of clinical responders at or beyond week 12, and the total number of clinical non-responders at or beyond week 12.

## 2.0 Data Analysis Considerations

## 2.1 Types of Analyses

Efficacy, safety, and descriptive analyses will be performed on the data collected in this trial.

## 2.2 Analysis Populations

The following analysis populations will be defined.

**Safety population** – The safety population includes all patients that have been enrolled in the study and injected with at least one dose of Tc 99m tilmanocept.

**Intent-to-diagnose (ITD) population** – Patients in the safety population meeting the following criteria are members of the ITD population:

- were injected with Tc 99m tilmanocept at Visit 2 (Day 0)
- received planar imaging of the hands at Visit 2 (Day 0)

This population will include all patients for whom a prediction might be made, although some patients may be excluded from analysis under this definition if a prediction cannot be made due to missing imaging or clinical data.

**Per-protocol (PP) population** – The PP population will include all ITD patients without major protocol violations. All protocol deviations will be classified as major or minor prior to database lock.

All efficacy analyses will be carried out on the ITD and PP populations with the ITD population being the primary analysis set. All analyses of safety data and baseline patient characteristics will be carried out on the safety population. A data listing displaying the patients excluded from each population will be created, as shown in Appendix B.

## 2.2.1 Subgroup Definitions and Considerations

Summaries of the agreement between the primary TUV prediction algorithm and all clinical outcomes will be performed in the following subgroups:

- Age (< 60 years, 60 years and older)</li>
- Sex
- Race (white, non-white)
- Time from RA diagnosis (< 5 years, 5 years and longer)
- Disease severity at baseline (moderate, severe)
- Previous use of biologics (yes, no)
- Previous and current use of DMARDs (background methotrexate only, other conventional DMARDs only, combination of methotrexate and other conventional DMARDs)
- Specific anti-TNFα therapy taken during trial
- Prednisone use on-study (on a stable dose, no prednisone use)
- ACPA level at baseline (high/low: 85 and above / < 85)</li>

The study will make every effort to enroll enough patients in each of these subgroups so that half-widths of the 95% confidence intervals of sensitivity and specificity are less than 20%. P-values on parameter estimates will not be included.

### 2.3 Missing Data Conventions

In the statistical analysis of the primary efficacy endpoints of the study, missing data will be handled according to the following table of missing data scenarios:

| Variable | Scenario | Primary Imputation Rule | Secondary<br>Imputation Rule |
|---|---|---|---|
| Clinical<br>Status at<br>Week 24 | Patient discontinued anti-TNFα therapy prior to Week 24 due to non- response to therapy | Patient classified as a clinical non-responder | N/A |

| Clinical<br>Status at<br>Week 24 | Patient discontinued study for reasons not attributable to non-response to therapy | Clinical status set to missing | Impute mean clinical response* |
|---|---|---|---|
| TUV<br>Prediction | Patient has TUV <sub>global[b]</sub> that is ≥ 5 but is missing week 5 imaging data | Impute mean prediction** | Prediction is Y (patient has improved) |
| TUV<br>Prediction | Patient is<br>missing<br>TUV <sub>global[b]</sub> | Prediction set to missing | N/A |

<sup>\*</sup>Mean clinical response will be calculated as follows: calculate the proportion of unique patients whose clinical status is Y (patient is a clinical responder), randomly allocate this proportion of "Y" to the missing clinical status at week 24 values. Assign all other missing clinical status values "N" (patient is clinical non-responder).

\*\*Mean prediction will be calculated as follows: using the patients for whom  $TUV_{global[b]} \geq 5$ , calculate the proportion whose TUV prediction is Y (patient has improved), randomly allocate this proportion of "Y" to the missing TUV predictions. Assign all other missing TUV predictions "N" (patient has not improved).

To assess the appropriateness of the missing data conventions for clinical status at week 24 and TUV prediction using mean imputation, tipping point analyses will be performed. Specifically, 95% confidence intervals for sensitivity and specificity will be plotted against increasing proportions of missing values imputed as "Y" to see at what point the conclusion of the study is reversed.

### 2.4 Interim Analyses

There are no interim analyses planned for this study.

#### 2.5 Calculation of TUV

TUV<sub>joint</sub> is defined to be the mean pixel intensity of the region of interest (ROI) defined by the reader divided by the mean pixel intensity of the hand reference region. Each of the three blinded readers will have determined the TUV distribution for both anterior and posterior views of the wrists and hands (wrists, MCPs, and PIPs) for the healthy patient normative data set. For all of the following calculations, the reader-specific TUV<sub>joint</sub> limits will be used. The upper

limit of normal is defined to be the upper limit of the 95% prediction interval of the joint-and-view-specific TUV in the normative data set.

For each RA patient do the following.

Step 1: Calculate TUV<sub>joint</sub> for each of the 22 DAS28 joints for which data are collected.

Step 2: Identify all imaged joints with TUV<sub>joint</sub> > upper limit of normal for the anatomically similar joint and view. These will be referred to as inflamed joints (IJ). Each joint has an anterior and posterior view: a joint is considered an IJ if either view has a TUV<sub>joint</sub> higher than the upper bound from the normative data set.

Step 3: Calculate the macrophage-involved contribution (MI) to Tc 99m tilmanocept localization for each IJ. This is done by expressing the TUV for the IJ as a fractional change from the mean TUV for the anatomically equivalent joint and view. That is, if TUV<sub>joint</sub> and  $\overline{\mathrm{H}}_{\mathrm{joint}}$  represent the joint and view specific TUV and the mean TUV for the anatomically equivalent joint and view from the normative data set respectively, the macrophage contribution to TUV is  $\mathrm{MI}_{\mathrm{joint}}$ :

$$MI_{joint} = \frac{TUV_{joint} - \overline{H}_{joint}}{\overline{H}_{joint}}.$$

Step 4:  $TUV_{global}$  is the total of the macrophage-involved contributions for the IJs. (Note that  $MI_k$  is effectively 0 if  $TUV_{joint}$  is less than or equal to the upper limit of normal from the normative data set.) That is,

$$TUV_{global} = \sum_{All\ IIs} MI_{IJ},$$

$$TUV_{global} = \sum_{k=1}^{22} MI_k.$$

The change in TUV<sub>global</sub> ( $\Delta$ TUV<sub>global[5w]</sub>) is the  $\Delta$ % from baseline:

$$\Delta TUV_{global[5w]} = 100 \cdot \frac{TUV_{global[5w]} - TUV_{global[b]}}{TUV_{global[b]}}.$$

## 2.6 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the control and supervision of the same Principal Investigator (PI). There will be no selective pooling of study centers.

#### 2.7 Documentation and Other Considerations

The data analyses will be conducted using SAS<sup>©</sup> Software, version 9.4 or later.

# 3.0 Analysis of Baseline Patient Characteristics

Baseline and demographic characteristics of the safety population (i.e., those injected with tilmanocept) will be summarized for all patients in the safety population. Continuous variables will be displayed via summary statistics (mean, median, sample size, standard deviation, minimum and maximum). Categorical variables will be summarized via counts and percentages.

Detailed listings of all baseline and demographic data for each patient will also be provided as shown in Section 7 below.

# 4.0 Analysis of Efficacy

# 4.1 Description of Efficacy Variables

## 4.1.1 Definition of Responder/Non-Responder Status

## **4.1.1.1 Prediction Algorithms**

The following two prediction algorithms will be defined for use in evaluating primary and secondary efficacy. Each algorithm will be used to predict a clinical response, and the subsequent prediction will be compared to the actual observed clinical response as described in Sections 4.1.2 and 4.1.3. In addition to these two prediction algorithms, the use of  $TUV_{global[b]}$  alone for the prediction of non-response will be analyzed as the key secondary efficacy variable. If  $TUV_{global[b]}$  is < 5 then the prediction is N (no improvement), otherwise, prediction is Y (improvement).

The  $\Delta TUV_{global[5w]}$  values will be used to predict improvement at 12 and 24 weeks according to algorithm 1. The  $\Delta TUV_{global[12w]}$  values will be used to predict improvement at 24 weeks according to algorithm 2. Both algorithms will be applied after the change in TUV calculations have been rounded to the nearest integer percentage (i.e., nearest hundredths place for a proportion).

## 1. ΔTUV<sub>global[5w]</sub> bucketing

In the below,  $TUV_{global}$  represents the global TUV at the current time point and  $TUV_{global[b]}$  represents the global TUV at baseline:

- If TUV<sub>global[b]</sub> is < 5 then the prediction is N (No improvement)
- Else if

$$\Delta TUV_{global[5w]} = \frac{TUV_{global[5w]} - TUV_{global[b]}}{TUV_{global[b]}} \le -0.10$$

the prediction is Y (patient has improved). That is, a patient will be predicted as improved if  $TUV_{global}$  goes down by greater than or equal to 10%.

Otherwise, the prediction is N.

#### 2. ∆TUV<sub>global[12w]</sub> bucketing

In the below, TUV<sub>global</sub> represents the global TUV at the current time point and TUV<sub>global[b]</sub> represents the global TUV at baseline:

- If TUV<sub>global[b]</sub> is < 5 then the prediction is N (No improvement)</li>
- Else if

$$\Delta TUV_{global[12w]} = \frac{TUV_{global[12w]} - TUV_{global[b]}}{TUV_{global[b]}} \leq -0.10$$

the prediction is Y (patient has improved). That is, a patient will be predicted as improved if  $TUV_{global}$  goes down by greater than or equal to 10%.

Otherwise, the prediction is N.

Tables which display the concordance between the predictions from each algorithm vs. clinical assessment will be provided. A listing showing which algorithms provide a prediction of improvement vs. no improvement, by patient, will also be provided.

#### 4.1.1.2 Clinical Assessments

ACR Response is derived through a combination of reductions from baseline in swollen or tender joint counts as well as improvement from baseline in at least 3 of the other parameters (patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant [ESR]). This study will evaluate the following three levels of ACR Response:

 ACR20: An ACR20 indicates that 20% improvement is observed in tender and swollen joint counts as well as 20% improvement in at least 3 of the other 5 criteria.

- ACR50: An ACR50 indicates that 50% improvement is observed in tender and swollen joint counts as well as 50% improvement in at least 3 of the other 5 criteria.
- ACR70: An ACR70 indicates that 70% improvement is observed in tender and swollen joint counts as well as 70% improvement in at least 3 of the other 5 criteria.

Each patient will be classified as a yes or a no for whether they meet each of the above ACR Response Criteria at each of the applicable post-baseline time points. Note that the above criteria are nested, such that if a patient is a yes for ACR70 at a given time point, then the patient is also a yes for ACR50 and ACR20 for that same time point.

A patient will be classified as improved on the CDAI depending on the baseline score as follows:

- If the baseline value is greater than 22, a reduction of more than 12 will be classified as improved. Otherwise, the patient is not improved.
- If the baseline value is between 10 and 22 (inclusive) a decrease of more than 6 will classified as improved. Otherwise, the patient is not improved.
- If the baseline value is less than 10, a decrease of more than 1 will be classified as improved. Otherwise the patient is not improved.

A patient will be classified as improved on the DAS28 with a score change of greater than 1.2.

A decrease of at least 0.22 in the HAQ-DI will be classified as improved. Otherwise, the patient is not improved on the HAQ-DI.

## 4.1.2 Description of Primary Efficacy Variables

The primary efficacy variables for determining clinical response are the response/non-response status at 24 weeks to new or changed anti-TNF $\alpha$  bDMARD therapy for rheumatoid arthritis based on the ACR50 criterion. The primary efficacy variables for determining the predicted response and non-response are  $\Delta TUV_{qlobal[5w]}$  bucketing.

The co-primary efficacy endpoints of the study are:

- Specificity of ΔTUV<sub>global[5w]</sub> bucketing with respect to ACR50 at week 24.
- Sensitivity of ΔTUV<sub>global[5w]</sub> bucketing with respect to ACR50 at week 24.

#### 4.1.3 Description of Key Secondary Efficacy Variables

The key secondary efficacy endpoint is:

NPV of TUV<sub>global[b]</sub> with respect to ACR50 at week 24.

## 4.1.4 Description of Secondary Efficacy Variables

The secondary efficacy predictor variables are the findings based on prediction algorithms 1 and 2, as described in Section 4.1.1.

The secondary efficacy response variables are:

- CDAI score at baseline (CDAI<sub>b</sub>), 12 (CDAI<sub>12w</sub>) and 24 weeks (CDAI<sub>24w</sub>)
- ACR Response Criteria (ACR20, ACR50, ACR70) at 12 and 24 weeks
- DAS28 Score at baseline, 12 weeks, and 24 weeks
- Constituent scores of the ACR Response Criteria at baseline, 12 weeks, and 24 weeks, including:
  - o TJC
  - o SJC
  - Patient assessment of global disease activity
  - o Rheumatologist assessment of global disease activity
  - o Patient assessment of pain
  - o Patient assessment of physical function
  - Acute-phase reactant value
- Constituent scores of the CDAI score at baseline, 12 weeks, and 24 weeks, including:
  - o TJC
  - o SJC
  - Patient Global Assessment
  - Physician Global Assessment

The secondary efficacy endpoints are as follows:

- Sensitivity and specificity of ΔTUV<sub>global[5w]</sub> bucketing with respect to ACR50 at week 12.
- NPV, PPV, and OA of ΔTUV<sub>global[5w]</sub> bucketing with respect to ACR50 at weeks 12 and 24.
- NPV of TUV<sub>global[b]</sub> with respect to ACR50 at week 12
- TUV<sub>global[b]</sub> and response to new anti-TNFα bDMARD therapy defined by the change from baseline (CFB) of CDAI to 12 ± 1 weeks and 24 ± 1 weeks (ΔCDAI<sub>12w</sub> and ΔCDAI<sub>24w</sub>, respectively), by the CFB of DAS28 to 12 ± 1 weeks and 24 ± 1 weeks (ΔDAS28<sub>12w</sub> and ΔDAS28<sub>24w</sub>,

- respectively) and by the CFB in each of the ACR Response Criteria components at  $12 \pm 1$  weeks and at  $24 \pm 1$  weeks.
- ΔTUV<sub>global[5w]</sub> bucketing and response to new anti-TNFα bDMARD therapy defined by the CFB of CDAI to 12 ± 1 weeks and 24 ± 1 weeks (ΔCDAI<sub>12w</sub> and ΔCDAI<sub>24w</sub>, respectively).
- Concordance of ΔTUV<sub>global[5w]</sub> bucketing with clinical criteria, including ACR Response Criteria, CDAI, DAS28, and HAQ-DI<sup>©</sup>. Concordance between the predicted response or non-response status and the clinical criteria will be evaluated using NPV, PPV, sensitivity, specificity, and OA.
- Concordance of ΔTUV<sub>global[12w]</sub> bucketing with clinical criteria, including ACR Response Criteria, CDAI, DAS28, and HAQ-DI<sup>©</sup>. Concordance between the improvement classifications and the clinical criteria will be evaluated using NPV, PPV, sensitivity, specificity, and OA.
- Response to new anti-TNFα bDMARD therapy defined by the CFB of CDAI to 12 ± 1 weeks and 24 ± 1 weeks (ΔCDAI<sub>12w</sub> and ΔCDAI<sub>24w</sub>, respectively).
- The correlation of ΔTUV<sub>global[5w]</sub> bucketing and response to new anti-TNFα bDMARD therapy from baseline to 24 ± 1 weeks defined by the changes from baseline in each of the ACR Response Criteria components.
- Constituent parameters of CDAI<sub>12w</sub>, CDAI<sub>24w</sub>, ΔCDAI<sub>12w</sub>, ΔCDAI<sub>24w</sub>, ACR Response Criteria at 12 and 24 weeks, including:
  - o TJC
  - o SJC
  - Patient assessment of global disease activity
  - Rheumatologist assessment of global disease activity
  - Patient assessment of pain
  - o Patient assessment of physical function
  - Acute-phase reactant value

### 4.2 Analysis of Efficacy Variables

Efficacy analyses will be conducted on the ITD and PP populations, with the ITD population serving as the primary analysis population.

## 4.2.1 Analysis of Primary Efficacy Variables

The co-primary efficacy variables will be summarized by reader in a 2 by 2 contingency table displaying the cell frequencies and marginal totals at 24 weeks. The specificity of  $\Delta TUV_{global[5w]}$  bucketing and the sensitivity of  $\Delta TUV_{global[5w]}$  bucketing will be calculated for each reader. The 95% exact (Clopper-Pearson) confidence intervals will be provided for each of these parameters. Observed significance levels (p-values) for the exact binomial tests of specificity of  $\Delta TUV_{global[5w]}$  bucketing greater than 0.8 and sensitivity of

 $\Delta TUV_{global[5w]}$  bucketing greater than 0.65 (see hypotheses specified in Section 1.3 above) will be provided.

Sensitivity and specificity are defined according to the following cross-tabulation:

| | Clinical Response | | |
|--------------------|-------------------|----------------|----------------|
| Predicted Response | Responder | Non-Responder | Total |
| Responder | Α | В | T <sub>1</sub> |
| Non-Responder | С | D | $T_2$ |
| Total | T <sub>3</sub> | T <sub>4</sub> | N |

Sensitivity =  $A/T_3$ . Specificity =  $D/T_4$ .

The above 2 by 2 contingency table will also be used to calculate the secondary efficacy endpoints of NPV, PPV, and OA as follows:

$$NPV = D/T_2$$
.  
 $PPV = A/T_1$ .  
 $OA = (A + D)/N$ .

## 4.2.2 Analysis of Key Secondary Efficacy Variables

NPV of TUV<sub>global[b]</sub> will be calculated for each reader. The 95% exact (Clopper-Pearson) confidence intervals will be provided. Observed significance levels (p-values) for the exact binomial tests of NPV of TUV<sub>global[b]</sub> greater than 0.7 will be provided.

## 4.2.3 Analysis of Secondary Efficacy Variables

All RA quantitative assessment variables (CDAI, ACR Response Criteria component scores, DAS28 score, and HAQ-DI) will be summarized by computing the mean, standard deviation, number of observations, minimum, median, and maximum for the observed values at each time point and for the change from baseline for values collected after Day 0. The ACR Response Criteria will be summarized with a frequency table of the highest ACR Response level (None, ACR20, ACR50, ACR70) attained by that patient at that time point. That is, a patient who satisfies ACR50 also satisfies ACR20 but will not appear in the frequency count for ACR20.

The qualitative assessments will be summarized in a 2 by 2 contingency table displaying the cell frequencies and marginal totals by reader as shown in section

4.2.1 above. The PPV and NPV of the predicted response will be calculated for each reader, as will the OA. In addition, 95% exact confidence intervals will be provided for each of these parameters. Observed significance levels (p-values) for the exact binomial (Clopper-Pearson) tests of PPV and NPV (see sections 1.3 and 4.2.1 above) will be provided for each reader. These tests will be based on PPV of the predicted response greater than 0.65, and NPV of the predicted response greater than 0.7.

Concordance of improvement classification for: 1)  $\Delta TUV_{global[5w]}$  bucketing and 2)  $\Delta TUV_{global[12w]}$  bucketing with clinical criteria (ACR Response, CDAI, DAS28, and HAQ-DI) will be analyzed as follows. Note that the concordance of  $\Delta TUV_{global[5w]}$  bucketing with ACR50 at 24 weeks is evaluated as co-primaries (sensitivity and specificity). For each of the RA improvement criteria, a cross-classification table will be provided. The PPV, NPV, sensitivity, specificity, and OA will be calculated and 95% exact (Clopper-Pearson) confidence intervals will be provided. Observed significance levels (p-values) for the exact binomial (Clopper-Pearson) tests for sensitivity and specificity will be provided for each reader.

Figures displaying the  $\Delta TUV_{global}$  by time point (5, 12, and 24 weeks) will be created to display the relationship between  $\Delta TUV_{global}$  over time with the corresponding clinical response assessment (ACR20/50/70, DAS28, and CDAI) at the given time point.

The Kendall rank correlation between  $\Delta TUV_{global[5w]}$  with  $\Delta CDAI_{12w}$  and  $\Delta CDAI_{24w}$  will be computed and a 95% confidence interval for its value will be computed using Fisher's Z-transformation. Similarly, the Kendall rank correlation between  $\Delta TUV_{global[5w]}$  with changes from baseline in DAS28 and in each of the ACR Response Criteria components at weeks 12 and 24 will be computed and a 95% confidence interval for its value will be computed using Fisher's Z-transformation. The marginal distributions of the variables will be characterized with the mean, standard deviation, and the number of data pairs.

The additive effect of either quantitative or qualitative assessment of Tc 99m tilmanocept imaging will be assessed with a generalized linear mixed model with the logit link function. The patient's response status will be used as the response variable. Fixed model terms for the quantitative and qualitative plus quantitative assessments will be used. The quantitative assessment will be based on  $\Delta TUV_{global[5w]}$  bucketing. Random terms will be fit for the subject and reader within subject using the variance component model. A table displaying the partial hypothesis tests (Type 3 test) for the fixed effects will be displayed.

# 5.0 Analysis of Safety

All safety analyses will be performed on the Safety Population.

The safety analysis variables are defined as follows:

- Adverse Events (AEs)
- Clinical Laboratory Tests (hematology, serum chemistry, urinalysis, RA panel)
- ECG Parameters
- Vital Signs

#### **Adverse Events**

Adverse events will be observed for each patient from signing of informed consent until termination from the study. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®). A treatment-emergent AE (TEAE) is defined as an AE whose start date is on or after the initial procedure date. Based on the coded terms, frequencies of each TEAE will be summarized by MedDRA® preferred term within system organ class (SOC), by severity grade, and by relationship to Tc 99m tilmanocept.

A summary of TEAEs will be constructed showing the following:

- Number of patients with at least one TEAE
- TEAEs by severity grade
- TEAE by relationship to Tc 99m tilmanocept
- TEAEs by relationship of TEAE to study procedure
- Number of patients with at least one treatment emergent serious adverse event

Treatment-emergent serious adverse events (TESAEs) will be tabulated by MedDRA® preferred term within SOC.

A by-patient AE data listing of all AEs including verbatim term, coded term, grade, and relation to study drug will be provided.

#### **Clinical Laboratory Tests**

Clinical laboratory tests will be performed at screening (baseline) and after the image acquisition on each imaging day (Visits 2, 4, 6, and 8). Only RA panel lab values and abnormal clinical laboratory values will be assessed for clinical significance as applicable. For each quantitative laboratory test, summary statistics (mean, standard deviation, median, range, n) on the raw as well as their changes from baseline will be presented by timepoint. A shift table will also be produced to show the changes in lab values over time relative to the normal ranges.

If multiple labs were performed at a given visit, then the latest results will be summarized in the analysis tables. All collected lab data will be listed.

#### **ECG Parameters**

ECGs will be performed within 30-minutes before and after injection. For each ECG parameter (heart rate, QRS, QT, PR, and QTcF), summary statistics (mean, standard deviation, median, range, n) on the raw as well as their changes from baseline will be presented by timepoint. A shift table will be provided to show changes in the qualitative assessment (abnormal or normal) from baseline (preinjection) to post-injection. The baseline value for each of the post-injection ECG parameters will be the corresponding pre-injection time point. All ECG data will be listed.

## **Vital Signs**

Vital signs will be performed at screening and within 30-minutes before and after injection. Height and weight will be measured only at screening and will be summarized as part of the baseline and demographic information. For each vital sign (respiration rate, systolic blood pressure, diastolic blood pressure, heart rate and temperature), summary statistics (mean, standard deviation, minimum, maximum, n) on the raw as well as their changes from baseline will be presented by timepoint. The baseline value for each of the post-injection vital sign parameters will be the corresponding pre-injection time point. If there are multiple vital signs taken at any time point, then the latest set of vital signs will be used for the analysis. All vital sign data will be listed.

# 6.0 Other Relevant Data Analyses/Summaries

#### **6.1 Patient Completion**

A table will be constructed with counts of screen failures and enrolled patients. Of those enrolled, counts and percentages of patients withdrawing from the study before study completion and the number completing the study will be displayed. For those patients that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. A data listing of all patient completion and withdrawal data will also be constructed.

#### 6.2 Physical Exam

Physical exams will be performed at screening. All physical exam data will be listed.

## **6.3 Study Drug Administration**

The volume, the calculated mass dose, and radioactivity of Tc 99m tilmanocept injected will be summarized. All study drug administration data will be listed.

## 6.4 RA Evaluation and Screening Physical Exam

Each RA patient will undergo a DAS28 evaluation during screening and at weeks 5, 12, and 24. The swollen and tender joints will be identified and documented during the physical examination. Results of all DAS28 evaluations will be listed.

#### **6.5 Concomitant Medications**

All prior and concomitant medications will be listed, as shown in Appendix B. A separate data listing will be created to show only those medications that were taken for RA.

# 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 1 | Patient Disposition | X | X |
| 2 | Demographics and Baseline Data Summary Statistics -<br>Continuous Variables (Safety Population) | Х | X |
| 3 | Demographics and Baseline Data Summary Statistics– Categorical Variables (Safety Population) | Х | Х |
| 4 | Summary of Study Drug Administration (Safety Population) | Х | Х |
| 5 | Summary of TUV by Study Day and DAS28 Joint (ITD population) | Х | Х |
| 6 | Summary of TUV by Study Day and DAS28 Joint (PP Population) | Х | |
| 7 | RA Status Summaries (ITD Population) | Х | Х |
| 8 | RA Status Summaries (PP Population) | Х | |
| 9 | ACR Response Classification by Time Point (ITD Population) | Х | Х |
| 10 | ACR Response Classification by Time Point (PP Population) | Х | |
| 11 | Concordance of TUV <sub>global[b]</sub> Alone and of ΔTUV <sub>global[5w]</sub> Bucketing and Week 12 Clinical Improvement Criteria (ITD Population) | X | Х |
| 12 | Concordance of TUV <sub>global[b]</sub> Alone and of ∆TUV <sub>global[5w]</sub> Bucketing and Week 12 Clinical Improvement Criteria (PP Population) | Х | |
| 13 | Concordance of TUV <sub>global[b]</sub> Alone and of ∆TUV <sub>global[5w]</sub> Bucketing and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 14 | Concordance of TUV <sub>global[b]</sub> Alone and of ∆TUV <sub>global[5w]</sub> Bucketing and Week 24 Clinical Improvement Criteria (PP Population) | X | |
| 15 | Concordance of ΔTUV <sub>global[12w]</sub> Bucketing and Week 24 Clinical Improvement Criteria (ITD Population) | Х | Х |
| 16 | Concordance of ΔTUV <sub>global[12w]</sub> Bucketing and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 17 | Concordance of ΔTUV <sub>global[5w]</sub> Bucketing and Week 12 Clinical Improvement Criteria in Subgroups (ITD Population) | Х | Х |
| 18 | Concordance of ΔTUV <sub>global[5w]</sub> Bucketing and Week 12 Clinical Improvement Criteria in Subgroups (PP Population) | Х | |
| 19 | Concordance of ΔTUV <sub>global[5w]</sub> Bucketing and Week 24 Clinical Improvement Criteria in Subgroups (ITD Population) | Х | |
| 20 | Concordance of ΔTUV <sub>global[5w]</sub> Bucketing and Week 24 Clinical Improvement Criteria in Subgroups (PP Population) | Х | |
| 21 | Concordance of Qualitative Assessment of Tc 99m Tilmanocept Imaging and Week 12 Clinical Improvement Criteria (ITD Population) | Х | Х |

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 22 | Concordance of Qualitative Assessment of Tc 99m Tilmanocept Imaging and Week 12 Clinical Improvement Criteria (PP Population) | X | В |
| 23 | Concordance of Qualitative Assessment of Tc 99m Tilmanocept Imaging and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 24 | Concordance of Qualitative Assessment of Tc 99m Tilmanocept Imaging and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 25 | Concordance of Qualitative plus Quantitative Assessment of Tc 99m Tilmanocept Imaging and Week 12 Clinical Improvement Criteria (ITD Population) | Х | |
| 26 | Concordance of Qualitative plus Quantitative Assessment of Tc 99m Tilmanocept Imaging and Week 12 Clinical Improvement Criteria (PP Population) | Х | |
| 27 | Concordance of Qualitative plus Quantitative Assessment of Tc 99m Tilmanocept Imaging and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 28 | Concordance of Qualitative plus Quantitative Assessment of Tc 99m Tilmanocept Imaging and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 29 | Kendall Rank Correlation of ΔTUV, ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 5 weeks (ITD Population) | Х | Х |
| 30 | Kendall Rank Correlation of ΔTUV, ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 5 weeks (PP Population) | Х | |
| 31 | Kendall Rank Correlation of ΔTUV, ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 12 weeks (ITD Population) | Х | Х |
| 32 | Kendall Rank Correlation of ΔTUV, ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 12 weeks (PP Population) | Х | |
| 33 | Kendall Rank Correlation of $\Delta$ CDAI, $\Delta$ ACR Response Criteria Components, and $\Delta$ DAS28 with $\Delta$ TUV at 24 weeks (ITD Population) | Х | Х |
| 34 | Kendall Rank Correlation of $\Delta$ CDAI, $\Delta$ ACR Response Criteria Components, and $\Delta$ DAS28 with $\Delta$ TUV at 24 weeks (PP Population) | Х | |
| 35 | Summary of Generalized Linear Mixed Model to Asses the Additive Effect of either Quantitative or Qualitative assessment of Tc 99m Tilmanocept Imaging on Patient Response Status at Week 12 (ITD Population) | Х | Х |
| 36 | Summary of Generalized Linear Mixed Model to Asses the Additive Effect of either Quantitative or Qualitative assessment of Tc 99m Tilmanocept Imaging on Patient Response Status at Week 12 (PP Population) | Х | |
| 37 | Summary of Generalized Linear Mixed Model to Asses the Additive Effect of either Quantitative or Qualitative assessment | Х | |

| Table<br>No. | Table Title | Included in Final Tables | Shown in Appendix B |
|---|---|---|---|
| | of Tc 99m Tilmanocept Imaging on Patient Response Status at Week 24 (ITD Population) | | |
| 38 | Summary of Generalized Linear Mixed Model to Asses the Additive Effect of either Quantitative or Qualitative assessment of Tc 99m Tilmanocept Imaging on Patient Response Status at Week 24 (PP Population) | Х | |
| 39 | Number and Percentage of Patients with TEAEs (Safety Population) | Х | Х |
| 40 | Summary of TEAEs (Safety Population) | Х | Х |
| 41 | Number and Percentage of Patients with TESAEs (Safety Population) | Х | Х |
| 42 | Number and Percentage of Patients with TEAEs by Severity Grade (Safety Population) | Х | Х |
| 43 | Number and Percentage of Patients with TEAEs by Level of Relationship to Tc 99m Tilmanocept (Safety Population) | Х | Х |
| 44 | Serum Chemistry Clinical Laboratory Parameters Summary Statistics (Safety Population) | Х | Х |
| 45 | Hematology Clinical Laboratory Parameters Summary Statistics (Safety Population) | Х | |
| 46 | Urinalysis Clinical Laboratory Parameters Summary Statistics (Safety Population) | Х | |
| 47 | Serum Chemistry Clinical Laboratory Parameters Shift Table (Safety Population) | Х | Х |
| 48 | Hematology Clinical Laboratory Parameters Shift Table (Safety Population) | Х | |
| 49 | Urinalysis Clinical Laboratory Parameters Shift Table (Safety Population) | Х | |
| 50 | ECG Parameters Summary Statistics (Safety Population) | Х | Х |
| 51 | ECG Shift Table (Safety Population) | Х | Х |
| 52 | Vital Signs Summary Statistics (Safety Population) | Х | Х |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Figures | Shown in<br>Appendix<br>B |
|---|---|---|---|
| Fig1 | Plot of $\Delta TUV_{global}$ by Imaging Time Point and ACR20 (ITD Population) | Х | Х |
| Fig2 | Plot of ΔTUV <sub>global</sub> by Imaging Time Point and ACR50 (ITD Population) | Х | |
| Fig3 | Plot of ΔTUV <sub>global</sub> by Imaging Time Point and ACR70 (ITD Population) | Х | |
| Fig4 | Plot of ΔTUV <sub>global</sub> by Imaging Time Point and CDAI (ITD Population) | Х | |
| Fig5 | Plot of ΔTUV <sub>global</sub> by Imaging Time Point and DAS28 (ITD Population) | Х | |
| Fig6 | Sensitivity Analysis #1 – Tipping Point Analysis to Assess the Appropriateness of Imputation of Clinical Status at Week 24 (ITD Population) | Х | Х |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Figures | Shown in Appendix B |
|---|---|---|---|
| Fig7 | Sensitivity Analysis #2 – Tipping Point Analysis to Assess the Appropriateness of Imputation of TUV Prediction (ITD Population) | X | |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix<br>B |
|---|---|---|---|
| DL1 | Patient Disposition Data Listing | Х | Х |
| DL2 | Inclusion/Exclusion Data Listing | Х | Х |
| DL3 | Protocol Deviations Data Listing | Х | Х |
| DL4 | Demographics Data Listing | Х | Х |
| DL5 | Patients Excluded from ITD Population Data Listing | Х | Х |
| DL6 | Patients Excluded from PP Population Data Listing | Х | Х |
| DL7 | Patients Excluded from Safety Population Data Listing | Х | Х |
| DL8 | Medical History Data Listing | Х | Х |
| DL9 | Prior and Concomitant Medications Data Listing | Х | Х |
| DL10 | Prior and Concomitant RA Medications Data Listing | Х | Х |
| DL11 | Adverse Events Data Listing | Х | Х |
| DL12 | Patient Laboratory Profiles – Hematology Data Listing | Х | Х |
| DL13 | Patient Laboratory Profiles – Serum Chemistry Data Listing | Х | |
| DL14 | Patient Laboratory Profiles – Urinalysis Data Listing | Х | |
| DL15 | Patient Laboratory Profiles – Rheumatology Panel Data<br>Listing | Х | |
| DL16 | Physical Exam Data Listing | Х | Х |
| DL17 | ACR/EULAR 2010 Classification Data Listing | Х | X |
| DL18 | ACR Data Listing | Х | Х |
| DL19 | CDAI, DAS28, HAQ-DI, and WPI Scores Data Listing | Х | Х |
| DL20 | DAS28 by Joint Data Listing | Х | Х |
| DL21 | DAS28 by Patient Data Listing | Х | Х |
| DL22 | Vital Signs Data Listing | Х | Х |
| DL23 | ECG Parameters Data Listing | Х | Х |
| DL24 | Study Drug Administration Data Listing | Х | Х |
| DL25 | Post-Injection Imaging Data Listing | Х | Х |
| DL26 | SPECT/CT Reader Results Data Listing – Hands and Wrists | Х | Х |
| DL27 | TUV Data Listing | Х | Х |
| DL28 | Qualitative Assessment Data Listing | Х | Х |
| DL29 | Qualitative plus Quantitative Assessments which differ from Original Quantitative Assessment | Х | Х |
| DL30 | ACR Response Criteria Data Listing | Х | Х |

# 8.0 References

N/A

## **Appendix A – Tables, Figures and Listing Specifications**

#### Orientation

Tables and figures will be displayed in landscape.

#### Margins

Margins will be 1 inch on all sides. Table and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### Headers

The table number will be on the first line of the title. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, 1 line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (Date)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

#### **Table Disclaimer**

The format of the mock tables shown in the appendix of this SAP will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

# **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

## **Display of Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (i.e., for a missing day value, the value displayed is in yyyy-mm format).

Statistical Analysis Plan Study No. NAV3-33

**Appendix B – Table, Figure, and Listing Shells**
Page x of y

Table 1. Patient Disposition
Navidea Biopharmaceuticals - Study No. NAV3-33

| | | | rerall<br>= xx) |
|-------------------|----------------------------------|----|-----------------|
| Screen Failures | | | XX |
| Enrolled | | | xx |
| Completed | | XX | (xxx%) |
| Withdrawn | | XX | (xxx%) |
| Withdrawal Reason | Adverse Event Protocol Violation | XX | (xxx%) |
| | Lost to Follow Up | XX | (xxx%) |
| | Withdrawal of Consent | XX | (xxx%) |
| | Sponsor Discretion | XX | (xxx%) |
| | Investigator Discretion | XX | (xxx%) |
| | Death | XX | (xxx%) |
| | Other | XX | (xxx%) |

The denominator for all percentages in the table is the number of enrolled patients. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 2. Demographics and Baseline Data Summary Statistics - Continuous Variables Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| Variable | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|
| Age (years) | XXX | xxx | xxx | XXX | xxx | XXX |
| Height (inches) | XXX | xxx | XXX | xxx | xxx | xxx |
| Weight (pounds) | xxx | xxx | xxx | xxx | XXX | xxx |
| Time from Diagnosis of RA (months) a | xxx | xxx | xxx | xxx | xxx | XXX |

<sup>&</sup>lt;sup>a</sup> Calculated as the difference between date of enrollment and date of RA diagnosis. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 3. Demographics and Baseline Data Summary Statistics - Categorical Variables
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | | Overall |
|---|---|---|
| Variable | Category | (N=xxx) |
| Gender | Male | xxx (xxx%) |
| | Female | xxx (xxx%) |
| Race | American Indian or Alaska Native | xxx (xxx%) |
| | Asian | xxx (xxx%) |
| | Black or African American | xxx (xxx%) |
| | Native Hawaiian or Other Pacific Islander | xxx (xxx%) |
| | White | xxx (xxx%) |
| | Other | |
| Ethnicity | Hispanic or Latino | xxx (xxx%) |
| | Not Hispanic or Latino | xxx (xxx%) |
| Severity of Disease | Mild | xxx (xxx%) |
| | Moderate | xxx (xxx%) |
| | Severe | xxx (xxx%) |
| Age Group | < 60 Years | xxx (xxx%) |
| | 60 Years and Older | xxx (xxx%) |
| Previous Use of Biologics | Yes | xxx (xxx%) |
| | No | xxx (xxx%) |
| Baseline ACPA Level | Low (< 85) | xxx (xxx%) |
| | High (85 and Above) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 4. Summary of Study Drug Administration Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|
| Tc 99m Dose (mCi) | xxxx | xxxx | xx | xxxx | xxxx | xxxx |
| Mass Dose (μg) | xxxx | xxxx | xx | xxxx | xxxx | xxxx |
| Total Volume of Tc 99m Tilmanocept Injected (mL) | xxxx | xxxx | xx | xxxx | xxxx | xxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 5. Summary of TUV by Study Day and DAS28 Joint
Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

| | | | Number | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| DAS28 Joint | Study Day | View | of Patients | Mean | Std Dev | n | Min | Max | Median | %CV |
| xxxxxxxxxxxx | XXXX | XXXXXXXX | XX | xxxx.x | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x | XXXX.X |
| | | XXXXXXXX | XX | xxxx.x | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | XXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | xxxx.x | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| xxxxxxxxxxxxxx | XXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | xxx | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | xxx | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | XXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | xxx | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | | xxxxxxxx | XX | xxxx.x | xxxx.x | xxx | xxxx.x | xxxx.x | xxxx.x | xxxx.x |
| xxxxxxxxxxxxxx | xxxx | xxxxxxxx | XX | xxxx.x | xxxx.x | xxx | xxxx.x | xxxx.x | xxxx.x | xxxx.x |
| | | xxxxxxxx | XX | xxxx.x | xxxx.x | xxx | xxxx.x | xxxx.x | xxxx.x | xxxx.x |
| | xxxx | xxxxxxxx | XX | xxxx.x | xxxx.x | XXX | xxxx.x | xxxx.x | xxxx.x | xxxx.x |
| | | xxxxxxxx | xx | xxxx.x | xxxx.x | xxx | xxxx.x | xxxx.x | xxxx.x | xxxx.x |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format is repeated for the PP population (table 6).

Page x of y

# Table 7. RA Status Summaries Navidea Biopharmaceuticals - Study No. NAV3-33 ITD Population (N=xxx)

| RA Status | Study | Data | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Measure | Visit | Type | Mean | Deviation | n | Min | Max | Median |
| XXXXXXXXXX | XXX | Baseline | XXXX.X | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| | XXX | RAW | xxxx.x | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | CFB | XXXX.X | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| XXXXXXXXXX | XXX | Baseline | xxxx.x | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| | XXX | RAW | XXXX.X | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | CFB | XXXX.X | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| XXXXXXXXXX | XXX | Baseline | xxxx.x | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| | XXX | RAW | XXXX.X | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | CFB | xxxx.x | XXX.XX | XXX | XXXX.X | XXXX.X | XXXX.X |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format is repeated for the PP population (table 8).

Page x of y

Table 9. ACR Response Classification by Time Point Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

| | Assessment | | | |
|---|---|---|---|---|
| Time Point | None | ACR20 | ACR50 | ACR70 |
| Week 5 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Week 12 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Week 24 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Table Format Repeats for PP Population (table 10).

Page x of y

Table 11. Concordance of  $TUV_{global[b]}$  Alone and of  $\Delta TUV_{global[5w]}$  Bucketing and Week 12 Clinical Improvement Criteria

Navidea Biopharmaceuticals - Study No. NAV3-33 ITD Population (N=xxx)

Part 1 of 6: ACR20

| | | | Clinical A | Assessment | | | |
|---|---|---|---|---|---|---|---|
| TUV Prediction | | Algorithm | | Not | = | | |
| Algorithm | Reader | Classification | Improved | Improved | Total | Measure | Value <sup>a</sup> |
| TUV <sub>global[b]</sub> Alone | х | Not Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | NPV<br>Confidence Limits<br>p-value | xxxx<br>(xxxx, xxxx)<br>x.xxxx |
| $\Delta \text{TUV}_{\text{global}[5w]}$ Bucketing | Х | Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Sensitivity<br>Confidence Limits<br>p-value | xxxx<br>(xxxx, xxxx)<br>x.xxxx |
| | | Not Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | - | |
| | | | | | | Specificity | XXXX |
| | | Total | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Confidence Limits | (xxxx, xxxx) |
| | | | | | | p-value | X.XXX |
| | | | | | | NPV Confidence Limits PPV Confidence Limits OA Confidence Limits | xxxx<br>(xxxx, xxxx)<br>xxxx<br>(xxxx, xxxx)<br>xxxx<br>(xxxx, xxxx) |

<sup>&</sup>lt;sup>a</sup> p-values of TUV Alone for NPV testing Ho:  $\pi$  = 0.7 and of TUV Bucketing for sensitivity testing Ho:  $\pi$  = 0.65 and specificity testing Ho:  $\pi$  = 0.8.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Within each part, the above two TUV prediction algorithm results will be displayed for each reader and sorting will be done by reader then prediction algorithm. For TUV Alone, the only reported outcome measure is NPV. For TUV Bucketing, outcome measures will include sensitivity, specificity, PPV, NPV, and OA, as shown above.

This format repeats for Part 2 (ACR50), Part 3 (ACR70), Part 4 (CDAI), Part 5 (DAS28), and Part 6 (HAQ-DI). Full table format repeats for PP population (table 12) and for tables 13 – 14.

Page x of y

Table 15. Concordance of  $\Delta TUV_{global[12w]}$  Bucketing and Week 24 Clinical Improvement Criteria Navidea Biopharmaceuticals - Study No. NAV3-33 ITD Population (N=xxx)

Part 1 of 6: ACR20

Clinical Assessment

| $\Delta exttt{TUV}_{	exttt{global}[12w]}$ Bucketing Classification | Improved | Not<br>Improved | Total | Measure | Value |
|---|---|---|---|---|---|
| Improved | vvv (vvv <sup>§</sup> ) | vvv (vvv%) | vvv (vvv%) | DDW | xxxx |
| Imploved | AAA (AAA®) | AAA (AAA®) | AAA (AAA®) | | (xxxx, xxxx) |
| Not Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Confidence Elmics | (AAAA, AAAA) |
| - | | | | NPV | xxxx |
| Total | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Confidence Limits | (xxxx, xxxx) |
| | | | | Sensitivity | XXXX |
| | | | | Confidence Limits | (xxxx, xxxx) |
| | | | | Specificity | xxxx |
| | | | | Confidence Limits | (xxxx, xxxx) |
| | | | | OA | xxxx |
| | | | | Confidence Limits | (xxxx, xxxx) |
| | Bucketing Classification Improved Not Improved | Bucketing Classification Improved Improved xxx (xxx%) Not Improved xxx (xxx%) | Bucketing Not Classification Improved Improved Improved xxx (xxx%) xxx (xxx%) Not Improved xxx (xxx%) xxx (xxx%) | Bucketing Not Classification Improved Improved Total Improved xxx (xxx%) xxx (xxx%) xxx (xxx%) Not Improved xxx (xxx%) xxx (xxx%) xxx (xxx%) | Bucketing |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Within each part, the above will be displayed for each reader. This format repeats for Part 2 (ACR50), Part 3 (ACR70), Part 4 (CDAI), Part 5 (DAS28), and Part 6 (HAQ-DI). Full table format repeats for PP population (table 16).

Page x of y

Table 17. Concordance of  $\Delta TUV_{global[5w]}$  Bucketing and Week 12 Clinical Improvement Criteria in Subgroups Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

Part 1 of 6: ACR20

| | | | Clinical A | Assessment | | | |
|---|---|---|---|---|---|---|---|
| Subgroup | Reader | $\Delta ext{TUV}_{	ext{global[5w]}}$ Bucketing Classification | Improved | Not<br>Improved | Total | Measure | Value |
| Female (N=xx) | х | Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | PPV<br>Confidence Limits | xxxx<br>(xxxx, xxxx) |
| | | Not Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | NPV<br>Confidence Limits | (xxxx (xxxx) |
| | | Total | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Sensitivity Confidence Limits Specificity Confidence Limits OA Confidence Limits | (XXXX) (XXXX, XXXX) XXXX (XXXX, XXXX) XXXX (XXXX, XXXX) |
| xxxxxxxxx (N=xx) | Х | Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | PPV | xxxx |
| | | Not Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Confidence Limits<br>NPV<br>Confidence Limits | (xxxx, xxxx)<br>xxxx<br>(xxxx, xxxx) |
| | | Total | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Sensitivity Confidence Limits Specificity Confidence Limits OA Confidence Limits | (XXXX<br>(XXXX, XXXX)<br>XXXX<br>(XXXX, XXXX)<br>XXXX<br>(XXXX, XXXX) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Within each part, the above will be displayed for each reader and subgroup, sorted by reader then subgroup. This format repeats for Part 2 (ACR50), Part 3 (ACR70), Part 4 (CDAI), Part 5 (DAS28), and Part 6 (HAQ-DI). Full table format repeats for PP population (table 18) and for tables 19 - 20.

Page x of y

Table 21. Concordance of Qualitative Assessment of Tc 99m Tilmanocept Imaging and Week 12 Clinical Improvement Criteria

Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

Part 1 of 6: ACR20

| | | Clinical | Assessment | | | |
|---|---|---|---|---|---|---|
| Reader | Qualitative<br>Assessment | Not<br>Improved Improved | | Total | Measure | Value <sup>a</sup> |
| Х | Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | PPV<br>Confidence Limits | xxxx<br>(xxxx, xxxx) |
| | Mak Turana d | | ( | ( | p-value | x.xxxx |
| | Not Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | NPV | xxxx |
| | Total | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Confidence Limits p-value | (xxxx, xxxx)<br>x.xxxx |
| | | | | | OA<br>Confidence Limits | xxxx<br>(xxxx, xxxx) |

Within each part, the above will be displayed for each reader. This format repeats for Part 2 (ACR50), Part 3 (ACR70), Part 4 (CDAI), Part 5 (DAS28), and Part 6 (HAQ-DI). Full table format repeats for PP population (table 22) and for tables 23 – 28.

 $<sup>^{\</sup>rm a}$  p-values for PPV testing Ho:  $\pi$  = 0.65 and for NPV testing Ho:  $\pi$  = 0.7. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 29. Kendall Rank Correlation of  $\Delta$ TUV,  $\Delta$ CDAI,  $\Delta$ ACR Response Criteria Components, and  $\Delta$ DAS28 with  $\Delta$ TUV at 5 Weeks

Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

Part 1 of 3: Reader x

| Measure <sup>a</sup> | Component<br>Parameter | Time Point | Kendall<br>Correlation <sup>b</sup> | 95% Confidence<br>Limits <sup>c</sup> | n | Mean | Standard<br>Deviation |
|---|---|---|---|---|---|---|---|
| ΔΤUV | | 5 Weeks | | | xxx | xxxxxx | xxxxxx |
| $\Delta$ TUV | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxx |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| $\Delta$ CDAI | Overall | 5 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | XXX | XXXXXX | xxxxxx |
| ΔCDAI | xxxxxxx | 5 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | XXXXXX | xxxxxx |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | XXX | XXXXXX | xxxxxx |
| ΔACR | xxxxxxx | 5 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | XXXXXX | xxxxxx |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | XXX | XXXXXX | xxxxxx |
| ΔDAS28 | | 5 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| | | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | XXXXXX | xxxxxx |

<sup>&</sup>lt;sup>a</sup> Change in ACR will be evaluated through the following components of the ACR Response Criteria: swollen joint count, tender joint count, patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant (ESR).

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format is repeated for each reader. Entire table (all parts) is repeated for the PP population (table 30).

 $<sup>^{</sup>m b}$  Kendall rank correlation between  $\Delta$ TUV at 5 weeks and the indicated measurement and time point.

<sup>&</sup>lt;sup>c</sup> Confidence limits calculated using Fisher's Z-transformation.

Page x of y

Table 31. Kendall Rank Correlation of  $\Delta$ TUV,  $\Delta$ CDAI,  $\Delta$ ACR Response Criteria Components, and  $\Delta$ DAS28 with  $\Delta$ TUV at 12 Weeks

Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

Part 1 of 3: Reader x

| | Component | | Kendall | 95% Confidence | | | Standard |
|---|---|---|---|---|---|---|---|
| Measurea | Parameter | Time Point | Correlation <sup>b</sup> | Limitsc | n | Mean | Deviation |
| ΔΤUV | | 12 Weeks | | | xxx | xxxxxx | xxxxxx |
| $\Delta$ TUV | | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxx | xxxxxx |
| $\Delta$ CDAI | Overall | 12 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | XXX | XXXXXX | XXXXXX |
| ΔCDAI | xxxxxxx | 12 Weeks<br>24 Weeks | x.xxx<br>x.xxx | (x.xxx, x.xxx)<br>(x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| $\Delta$ ACR | xxxxxxx | 12 Weeks<br>24 Weeks | x.xxx<br>x.xxx | (x.xxx, x.xxx)<br>(x.xxx, x.xxx) | xxx<br>xxx | xxxxxx | xxxxxx |
| ΔDAS28 | | 12 Weeks<br>24 Weeks | x.xxx<br>x.xxx | (x.xxx, x.xxx)<br>(x.xxx, x.xxx) | xxx | xxxxxx | xxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format is repeated for each reader. Entire table (all parts) is repeated for the PP population (table 32).

<sup>&</sup>lt;sup>a</sup> Change in ACR will be evaluated through the following components of the ACR Response Criteria: swollen joint count, tender joint count, patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant (ESR).

 $<sup>^{</sup>m b}$  Kendall rank correlation between  $\Delta {
m TUV}$  at 12 weeks and the indicated measurement and time point.

<sup>&</sup>lt;sup>c</sup> Confidence limits calculated using Fisher's Z-transformation.

Page x of y

Table 33. Kendall Rank Correlation of  $\Delta$ CDAI,  $\Delta$ ACR Response Criteria Components, and  $\Delta$ DAS28 with  $\Delta$ TUV at 24 Weeks

Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

Part 1 of 3: Reader x

| Measurea | Component<br>Parameter | Time Point | Kendall<br>Correlation <sup>b</sup> | 95% Confidence<br>Limits <sup>c</sup> | n | Mean | Standard<br>Deviation |
|---|---|---|---|---|---|---|---|
| $\Delta$ TUV | | 24 Weeks | | | xxx | xxxxxx | xxxxxx |
| $\Delta$ CDAI | Overall | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxx | xxxxx |
| $\Delta$ CDAI | xxxxxxx | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxx | xxxxx |
| $\Delta$ ACR | xxxxxxx | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxx | xxxxx |
| ΔDAS28 | | 24 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format is repeated for each reader. Entire table (all parts) is repeated for the PP population (table 34).

<sup>&</sup>lt;sup>a</sup> Change in ACR will be evaluated through the following components of the ACR Response Criteria: swollen joint count, tender joint count, patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant (ESR).

 $<sup>^{</sup>m b}$  Kendall rank correlation between  $\Delta$ TUV at 24 weeks and the indicated measurement and time point.

 $<sup>^{\</sup>mbox{\tiny c}}$  Confidence limits calculated using Fisher's Z-transformation.

Table 35. Summary of Generalized Linear Mixed Model to Asses the Additive Effect of either Quantitative or Qualitative Assessment of Tc 99m Tilmanocept Imaging on Patient Response Status at Week 12

Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

| Model Term <sup>a</sup> | Parameter<br>Estimate <sup>b</sup> | Standard Error | 95% Confidence<br>Limits | p-value° |
|---|---|---|---|---|
| 110001 101111 | 2001 | 204114414 21101 | 21111200 | P varao |
| Quantitative Imaging<br>Assessment | xxx.xxx | xxx.xxx | (xxx.xxx, xxx.xxx) | x.xxx |
| Qualitative plus<br>Quantitative Imaging<br>Assessment | xxx.xxx | xxx.xxx | (xxx.xxx, xxx.xxx) | x.xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table is repeated for the PP population (table 36) and for tables 37 – 38.

Page x of y

a Indicator variable for prediction of "Improved" compared to the reference category of "Not Improved."

<sup>&</sup>lt;sup>b</sup> Estimate calculated from a generalized linear mixed model with the logit link function with patient response status as the response variable, fixed terms for quantitative and qualitative plus quantitative imaging assessment, and random terms for subject and reader within subject using a variance component model.

 $<sup>^{\</sup>circ}$  Based on a two-sided t-test.

Table 39. Number and Percentage of Patients with TEAEs
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | Overall |
|---------------------------------|------------|
| Adverse Event Categorya: | (N=xxx) |
| Total Number of TEAEs | xxx |
| Patients with at Least One TEAE | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

## Table 40. Summary of TEAEs Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| | Overall (N=xxx) |
|---|---|
| Patients With at Least One TEAE | xxx |
| Maximum TEAE Severity Grade | |
| Mild | xxx (xxx%) |
| Moderate | xxx (xxx%) |
| Severe | xxx (xxx%) |
| Highest Relationship of TEAE to Tc 99m tilmanocept Definitely Not [n(%)] Probably Not [n(%)] Possibly [n(%)] Probably [n(%)] Definitely [n(%)] | xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) |
| <pre>Highest Relationship of TEAE to Study Procedure Definitely Not [n(%)] Probably Not [n(%)] Possibly [n(%)] Probably [n(%)] Definitely [n(%)]</pre> | xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) |
| Patients with at Least One TESAE | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 41. Number and Percentage of Patients with TESAEs Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| Adverse Event Categorya: | Overall (N=xxx) |
|---|---|
| Total Number of TESAEs | xxx |
| Patients with at Least One TESAE | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 42. Number and Percentage of Patients with TEAEs by Severity Grade
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | | Severity Grad | de |
|---------------------------------|------------|---------------|------------|
| Adverse Event Categorya: | Mild | Moderate | Severe |
| Total Number of TEAEs | xxx | xxx | xxx |
| Patients with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | , , | , | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 43. Number and Percentage of Patients with TEAEs by Level of Relationship to Tc 99m Tilmanocept
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

Level of Relationship

| | | | | = | |
|---|---|---|---|---|---|
| | Definitely | Probably | Possibly | Probably | Definitely |
| Adverse Event Categorya: | Not | Not | Related | Related | Related |
| Total Number of TEAEs | XXX | XXX | XXX | XXX | XXX |
| Patients with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 44. Serum Chemistry Clinical Laboratory Parameters Summary Statistics
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|
| Parameter(units) | Visit | Data Typeª | Mean | Dev | n | Min | Max | Median |
| xxxxxxxx (xxx) | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | xxx | XXX | XXX | XXX | XXX | XXX |
| | Day 8 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| xxxxxxxx (xxx) | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | xxx | XXX |
| | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | xxx | XXX | XXX | XXX | XXX | XXX |
| | Day 8 | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | CFB | xxx | XXX | XXX | XXX | XXX | XXX |

Table format repeats for tables 45 and 46.

<sup>&</sup>lt;sup>a</sup> RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value). STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxxx.sas

Page x of y

Table 47. Serum Chemistry Clinical Laboratory Parameters Shift Table
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

Part 1 of 4: Day 0

#### Baseline Result/ Post-Injection Result

| Panel/Parameter (units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

### Table 47. Serum Chemistry Clinical Laboratory Parameters Shift Table Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

Part 2 of 4: Week 5

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 47. Serum Chemistry Clinical Laboratory Parameters Shift Table
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

Part 3 of 4: Week 12

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx(xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 47. Serum Chemistry Clinical Laboratory Parameters Shift Table
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

Part 4 of 4: Week 24

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx(xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 50. ECG Parameters Summary Statistics
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| ECG | | Data | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Parameter(units) | Visit | Typea | Mean | Std Dev | n | Min | Max | Median |
| xxxxxxxx (xxx) | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 5 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 5 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 12 Pre-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | (Baseline) | | | | | | | |
| | Week 12 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 24 Pre-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | (Baseline) | | | | | | | |
| | Week 24 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | xxx | XXX | XXX | XXX | XXX | xxx |

<sup>&</sup>lt;sup>a</sup> RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value). STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxxx.sas

Page x of y

Table 51. ECG Shift Table
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

Baseline Result/
Post-Injection Result

| Visit | Abnormal/<br>Abnormal | Abnormal/<br>Normal | Normal/<br>Abnormal | Normal/<br>Normal |
|---|---|---|---|---|
| xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| XXXXX | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| XXXXX | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 52. Vital Signs Summary Statistics
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| Vital Sign | | Data | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Parameter (units) | Visit | Typea | Mean | Std Dev | n | Min | Max | Median |
| xxxxxxxxx (xxx) | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 5 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 5 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 12 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 12 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Week 24 Pre-Injection(Baseline) | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | Week 24 Post-Injection | RAW | xxx | XXX | XXX | XXX | XXX | xxx |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

a RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value).

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Figure 1. Plot of  $\Delta TUV_{global}$  by Imaging Time Point and ACR20 Navidea Biopharmaceuticals - Study No. NAV3-33 ITD Population (N=xxx)

Part 1 of 3: Reader x



Responder status based on ACR20 at each week. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Figure format repeats for each part and for Figures 2-5. Footnote text will be updated in each figure to correspond to the clinical assessment noted in the title (ACR50, ACR70, CDAI, or DAS28).

Page x of y

Figure 6. Sensitivity Analysis #1 - Tipping Point Analysis to Assess the Appropriateness of Imputation of

Clinical Status at Week 24

Navidea Biopharmaceuticals - Study No. NAV3-33

ITD Population (N=xxx)

Part 1 or 2: Sensitivity



Remaining missing week 24 clinical status outcomes imputed as non-responders. Solid horizontal line represents 65% sensitivity. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Figure 6. Sensitivity Analysis #1 - Tipping Point Analysis to Assess the Appropriateness of Imputation of
Clinical Status at Week 24
Navidea Biopharmaceuticals - Study No. NAV3-33
ITD Population (N=xxx)

Part 2 of 2: Specificity



Remaining missing week 24 clinical status outcomes imputed as non-responders. Solid horizontal line represents 80% specificity. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Figure format repeats for Figure 7.

Page x of y

Data Listing 1. Patient Disposition Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33

| Patient<br>No. | Disposition Status | Date of<br>Completion or<br>Withdrawal | Withdrawal Reason |
|---|---|---|---|
| xxxx | *************************************** | xxxxxxxx | *************************************** |
| XXXX | xxxxxxxxxxxxxxxx | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | ************************************** |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 2. Inclusion/Exclusion Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33

| Patient<br>No. | Did Patient<br>Meet All<br>Eligibility<br>Criteria? | Criterion Category | Criterion | Was a<br>Waiver<br>Granted? | Is Patient a<br>Screen<br>Failure? |
|---|---|---|---|---|---|
| | | | | | _ |
| Xxxx | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | XXXX | XXXX |
| XXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |
| XXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | XXXX | XXXX |
| XXXX | xxxx | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx | XXXX | xxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 3. Protocol Deviations Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33

| Patient<br>No. | Date of<br>Deviation | Deviation Description | Deviation Category<br>(Major/Minor) |
|---|---|---|---|
| xxxx | xxxxxx | ******* | xxxxxxxxx |
| XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX |
| XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 4. Demographics Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| Patient<br>No. | Informed<br>Consent<br>Date/Time | Time from Diagnosis of RA (months) | Disease<br>Severity | Date<br>of<br>Birth | Height<br>(inches) | Weight<br>(pounds) | Age<br>(years) | Gender | Race | Ethnicity | Previous<br>Use of<br>Biologics<br>(Y/N) | Baseline<br>ACPA Level<br>(Low/High) <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxxxx | xxx | xxxxxx | xxxxxx | xxx | xxx | xxx | xxxxxx | xxxxxx | xxxxxx | Х | XXX |
| XXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | X | XXX |
| XXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | X | XXX |
| XXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | X | XXX |

<sup>&</sup>lt;sup>a</sup> Calculated as the difference between date of enrollment and date of RA diagnosis.

 $<sup>^{\</sup>rm b}$  Low is < 85, and High is 85 and above. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 5. Patients Excluded from ITD Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
All Enrolled Patients (N=xxx)

| Patient No. | Reason for Exclusion |
|-------------|----------------------------|
| XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| xxxx | XXXXXXXXXXXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas
Page x of y

Data Listing 6. Patients Excluded from PP Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
All Enrolled Patients (N=xxx)

| _ | Patient No. | Reason for Exclusion |
|---|-------------|-----------------------------|
| | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX |

Page x of y

Data Listing 7. Patients Excluded from Safety Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
All Enrolled Patients (N=xxx)

| Patient No. | Reason for Exclusion |
|-------------|--------------------------|
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |

Page x of y

Data Listing 8. Medical History Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | MedDRA System Organ Classa/ | | | |
|---|---|---|---|---|
| Patient | MedDRA Preferred Term/ | | Resolution/Stop | o<br>O |
| No. | CRF Verbatim Term | Start Date | Date | Ongoing? |
| Xxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |

<sup>&</sup>lt;sup>a</sup> Medical history terms coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

# Data Listing 9. Prior and Concomitant Medications Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

Drug Preferred Terma/

| | Verbatim/ | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Patient | ATC Level 1 Text/ | Prior | | | Start | Stop | | |
| No. | ATC Level 4 Text | Medication? | Indication | Frequency | Date | Date | Route | Ongoing? |
| Xxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxx | X | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 10. Prior and Concomitant RA Medications Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

Drug Preferred Terma/

| | Verbatim/ | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Patient | ATC Level 1 Text/ | Prior | | | Start | Stop | | |
| No. | ATC Level 4 Text | Medication? | Indication | Frequency | Date | Date | Route | Ongoing? |
| Xxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxx | X | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | | |

Medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 11. Adverse Events Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | | Start Date | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Start | and Time of | | MedDRA System Organ | | | | |
| | Date and | Nearest | | Class <sup>a</sup> / | | Relation to | | |
| | Time/ | Previous | | MedDRA Preferred | | Tc 99m | | |
| Patient | End Date | tilmanocept | Treatment | Term/ | | tilmanocept/ | | |
| No. | and Time | Injection | Emergent? | CRF Verbatim Term | Severity | Procedure | Serious? | Outcome |
| XXXXXXXX | XXXXXXX | XXXXXXX | XXX | xxxxxxxxxxxxxxx | xxxxxxx | xxxxxxxx/ | XXX | xxxxxxx |
| | xxxxxxx/ | XXXXXXX | | xxxxxxxxxxxxxxx | | XXXXXXX | | |
| | XXXXXXX | | | xxxxxxxxxxxxxx | | | | |
| | XXXXXXX | | | | | | | |
| XXXXXXXX | XXXXXXX | XXXXXXX | XXX | xxxxxxxxxxxxxx | XXXXXXX | xxxxxxxx/ | XXX | XXXXXXX |
| | xxxxxxx/ | XXXXXXX | | xxxxxxxxxxxxxx | | XXXXXXX | | |
| | XXXXXXX | | | xxxxxxxxxxxxxx | | | | |
| | XXXXXXX | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 12. Patient Laboratory Profiles - Hematology Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | | | | | Normal | l Range | |
|---|---|---|---|---|---|---|---|
| Patient | | Sample Date | | | | | = |
| No. | Visit | and Time | Lab Parameter (Units) | Result | Lab Low | Lab High | Clin. Sig? |
| XXXX | XXXXXXX | xxxxxxxx / xx:xx | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Table format is repeated for Serum Chemistry, Urinalysis, and Rheumatology Panel Listings (Listings 13, 14, 15).

Page x of y

Data Listing 16. Physical Exam Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| Patient | | Date | | | |
|---|---|---|---|---|---|
| No. | Visit | Conducted | Body System | Result | Abnormality |
| • | | | | | |
| XXXX | XXXXXXX | XXXXXXX | General Appearance | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Skin | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Eyes, Ears, Nose, Throat | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Head and Neck | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Lungs | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Heart | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Abdomen | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Lymph Nodes | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Musculoskeletal | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Nervous System | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Other: XXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page  ${\tt x}$  of  ${\tt y}$ 

Data Listing 17. ACR/EULAR 2010 Classification Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

### ACR/EULAR 2010

| Patient<br>No. | Visit | Date | Joint<br>Involvement | Serology | Acute-<br>Phase<br>Reactants | Duration<br>of<br>Symptoms | Total Score |
|---|---|---|---|---|---|---|---|
| xxxx | xxxxxxx | xxxxxxx | xxx | xxx | xxx | xxx | xxx |
| XXXX | xxxxxx | xxxxxx | xxx | xxx | xxx | xxx | xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

# Data Listing 18. ACR Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

ACR Components

| Patient | | | Tender<br>Joint | Swollen<br>Joint | Patient's<br>Global<br>Disease | Physician's<br>Global<br>Disease | Patient<br>Assessment | Patient<br>Assessment<br>Physical | Acute<br>Phase<br>Reactant | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | Visit | Date | Count | Count | Activity | Activity | of Pain | Function | Value | ACR20 | ACR50 | ACR70 |
| xxxx | xxxxxx | xxxxxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx |
| XXXX | XXXXXXX | XXXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Page x of y

Data Listing 19. CDAI, DAS28, HAQ-DI, and WPI Scores Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | | | | CDAI | Component | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Patient's | Physician's | | | | | HAQ- | |
| | | | Tender | Swollen | Global | Global | CDAI | | DAS28 | | DI | WPI |
| Patient | | | Joint | Joint | Disease | Disease | Total | CDAI | Total | DAS28 | Total | Total |
| No. | Visit | Date | Score | Score | Activity | Activity | Score | Improved | Score | Improved | Score | Score |
| XXXX | XXXXXXX | XXXXXXX | XXX | XXX | XXX | XXX | XXX | X | XX.X | X | XX.X | XX.X |
| xxxx | xxxxxxx | xxxxxxx | xxx | xxx | xxx | xxx | xxx | x | xx.x | x | xx.x | xx.x |

Page x of y

Data Listing 20. DAS28 by Joint Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

### DAS28 Joint Classification

| Patient | | | | Result | Result |
|---------|---------|---------|----------|--------------|-------------|
| No. | Visit | Date | Joint | (Right Body) | (Left Body) |
| XXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| XXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |

Page x of y

Data Listing 21. DAS28 by Patient Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| | | | | | DAS28 | | |
|---|---|---|---|---|---|---|---|
| | | • | | | Patient | Erythrocyte | |
| | | | Tender | Swollen | VAS | Sedimentation | |
| Patient | | | Joint | Joint | Global | Rate (ESR; | DAS28 |
| No. | Visit | Date | Count | Count | (mm) | mm/hr) | Score |
| xxxx | xxxxxx | xxxxxx | xxx | xxx | xxx | xxx | XXX |
| XXXX | xxxxxx | xxxxxx | XXX | xxx | xxx | xxx | XXX |

Page x of y

Data Listing 22. Vital Signs Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| | | | | | Systolic | Diastolic | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | Blood | Blood | Heart | |
| Patient | | | | Temp. | Pressure | Pressure | Rate | Respirations |
| No. | Visit | Date | Time | (°F) | (mmHg) | (mmHg) | (mqd) | per Minute |
| XXXX | XXXXXX | XXXXXXX | XXXXX | XXX | XXX | XXX | XXX | XXX |
| | | | XXXXX | XXX | XXX | XXX | XXX | XXX |
| | | | XXXXX | XXX | XXX | XXX | XXX | XXX |
| XXXX | XXXXXXX | XXXXXXX | XXXXX | XXX | XXX | XXX | XXX | XXX |
| | | | XXXXX | XXX | XXX | XXX | XXX | XXX |
| | | | XXXXX | XXX | XXX | XXX | XXX | XXX |

Page x of y

Data Listing 23. ECG Parameters Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| Patient<br>No. | Visit | Date | Time | Heart Rate (bpm) | PR Interval (msec) | QRS<br>Interval<br>(msec) | QT Interval (msec) | QTcF<br>Interval<br>(msec) | Overall<br>Interpretation |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxxxx | xxxxx | xxxxxx | xxxxxx | xxxxxxx | xxxxxxx | xxxxxx | xxxx | xxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Data Listing 24. Study Drug Administration Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| Patient<br>No. | Date/<br>Time of<br>Injection | Anatomic<br>Location<br>of<br>Injection | Pre-Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Post-<br>Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Calculated Amount of Administered Radioactivity (mCi) | Calculated<br>Mass Dose<br>(µg) | Volume<br>Injected<br>(mL) | Lot<br>Number |
|---|---|---|---|---|---|---|---|---|
| xxxx | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | xxx |
| XXXX | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | XXX | XXX | xxx |
| | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 25. Post-Injection Imaging Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| Patient<br>No. | Visit | Date of<br>Imaging | Start Time of Imaging | SPECT/CT Image<br>Finding |
|---|---|---|---|---|
| xxxx | xxxxxxx | xxxxxx | xx:xx | xxx |
| xxxx | xxxxxxxx | xxxxxx | xx:xx | XXX |

Page x of y

Data Listing 26. SPECT/CT Reader Results Data Listing - Hands and Wrists Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| Patient | Post-Injection | | SPECT/CT |
|---------|--------------------|-------------|---------------|
| No. | Imaging Time Point | Joint | Image Finding |
| , | | | |
| XXXX | XXXXXX | XXXXXXXXXXX | XXXX |
| | | XXXXXXXXXXX | |
| XXXX | XXXXXX | XXXXXXXXXXX | XXXX |
| | | ××××××××××× | |

Page x of y

## Data Listing 27. TUV Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

TUV Classification of Improvement

| Patient No. | Reader No. | Algorithms<br>Predicting<br>Improvement <sup>a</sup> | Algorithms<br>Predicting No<br>Improvement <sup>a</sup> | Visit | Date/Time | Region of<br>Interest <sup>b</sup> | TUV |
|---|---|---|---|---|---|---|---|
| XXXX | X | х, х | Х | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| | | | | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| | | | | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| | | | | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| | | | | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| xxxx | X | Х | X, X | xxxxxxx | xxxxxx | xxxxxx | XXXXX |

a 1 = Change in Global TUV[5w] Bucketing, 2 = Change in Global TUV[12w] Bucketing

b Region of Interest is joint or Global. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 28. Qualitative Assessment Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-33
Safety Population (N=xxx)

| Patient No. | Reader No. | Qualitative<br>Assessment <sup>a</sup> | Date/Time |
|---|---|---|---|
| xxxx | Х | xxxxxx | xxxxxxx/ |
| xxxx | Х | xxxxxxx | xxxx<br>xxxxxxxx/<br>xxxx |

<sup>&</sup>lt;sup>a</sup> Qualitative Assessment is either "Improved" or "Not Improved." STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 29. Qualitative plus Quantitative Assessments which differ from Original Quantitative

Assessment

Assessment Navidae Pierbergesentianla (Chudu Na. NAV. 22)

Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| Patient No. | Reader No. | Qualitative<br>plus<br>Quantitative<br>Assessment <sup>a</sup> | Date/Time of<br>Qualitative plus<br>Quantitative<br>Assessment | Original<br>Quantitative<br>Assessment <sup>a</sup> | Date/Time of<br>Original<br>Quantitative<br>Assessment |
|---|---|---|---|---|---|
| xxxx | х | xxxxxxx | xxxxxxx/ | xxxxxx | xxxxxxxx/ |
| xxxx | х | xxxxxxx | xxxx<br>xxxxxxxx/ | xxxxxx | xxxx<br>xxxxxxxx/ |

<sup>&</sup>lt;sup>a</sup> Assessment is either "Improved" or "Not Improved." STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

## Data Listing 30. ACR Response Criteria Data Listing Navidea Biopharmaceuticals - Study No. NAV3-33 Safety Population (N=xxx)

| Patient<br>No. | Visit | Highest ACR<br>Response<br>Assessment <sup>a</sup> | Number of<br>Tender<br>Joints | Number of<br>Swollen<br>Joints | Patient<br>Global<br>Assessment | Physician<br>Global<br>Assessment | HAQ Total | VAS Pain<br>Score | ESR |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxxxx | xxxxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx |
| xxxx | xxxxxx | xxxxx | XXX | xxx | xxx | XXX | xxx | xxx | xxx |

<sup>&</sup>lt;sup>a</sup> Options are None, ACR20, ACR50, or ACR70. Response assessment will be blank for baseline measurements. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas